CLINICAL TRIAL: NCT01378000
Title: Study Effects of Ultra-slow Continuous Intravenous Infusion of Unfractionated Heparin on Progressive Cerebral Infarction - a Clinical Study
Brief Title: Study on Continuous Intravenous of Unfractionated Heparin (UFH) to Treat Progressive Cerebral Infarction
Acronym: UHPCI
Status: Completed | Type: Observational
Sponsor: Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2010CZTCWM
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2010-09

CONDITIONS: Heparin Causing Adverse Effects in Therapeutic Use; Heparin-induced Thrombosis; Acute Cerebral Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- UFH,once a day
- heparin Calcium,every 12 hours
- dextran,Salviae,once a day
- UFH,continuous intravenous infusion,

SUMMARY:
A clinical trial to study the effects of dosage, infusion methods and complications of unfractionated heparin (UFH) treating acute progressive cerebral infraction was conducted. In this study, we observed the effects of four UFH treatments on 480 acute progressive cerebral infraction patients during from the 6th and the 72nd hour after the attack. It was concluded that the ultra-slow continuous intravenous infusion of UFH can significantly reduce the neurological deficit score of patients with progressive cerebral infarction, increase the cure rate, decrease the recurrence rate, and improve long-term quality of daily life. It is more effective than the treatment of intravenous infusion of low- molecular- weight UFH at once a day, and the risk of bleeding may not necessarily be increased.

DETAILED DESCRIPTION:
Treatment' effectiveness rates of the four groups were 95.80%, 85.22%, 85.47%, and 87.72% respectively. The result of Group A was significantly different from those of Group B, C, and D (p <0.05). The adverse complication occurrence rates of the four groups were 5.88%, 3.48%, 4.27% and 3.51%.

ELIGIBILITY:
Inclusion Criteria:

* Time after breakout: 6- 72 hours
* Blood pressure: below 180/100 mm Hg (1 mm Hg= 0.133 kPa)
* Paralyzed limb muscle strength: Level 0
* Being conscious or in mild or moderate coma, and hernia- free
* The nerve function continued to aggravate from several hours to a week after the breakout.
* No abnormal blood coagulation Platelet count Plt >10×109/L
* Brain CT or MRI confirming and ruling out the occurrence of bleeding
* Match the diagnostic standards of acute cerebral infraction established by the 4th Chinese China Neurology Association
* Informed consent Agreement Signed

Exclusion Criteria:

* History of intracranial hemorrhage bleeding risk or Plt <10 × 109/ L
* Record of severe heart, liver, or renal insufficiency or severe diabetes mellitus
* Infarct area larger than 1/3 of hemispheric area
* Pregnant

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From May 2003 to October 2009 480 patients of acute progressive cerebral infraction that matched the standards above were included in the research.
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
change of NIHSS at 4 weeks | 4 weeks
  the ultra-slow continuous intravenous infusion of UFH can significantly reduce the neurological deficit score of patients with progressive cerebral infarction,

SECONDARY OUTCOMES:
the recurrence rate at 6 months | 6 months
  the ultra-slow continuous intravenous infusion of UFH can significantly decrease the recurrence rate of patients with progressive cerebral infarction,
changs of ADL after 6 months | 6 months
  the ultra-slow continuous intravenous infusion of UFH can significantly improve ADL of patients with progressive cerebral infarction
Number of patients with Adverse Events | 4 weeks
  The adverse complication occurrence rates of the four groups have no significantly different

CONTACTS AND LOCATIONS:
Overall Officials: wang zh yong, professor, Principal Investigator — cangzhou hospital
Locations (1):
- Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei, China

REFERENCES:
- See also: cangzhou hospital — http://www.cz96130.com